CLINICAL TRIAL: NCT06319170
Title: A Multi-center, Open-label, Randomized, Parallel-group Trial to Characterize the Pharmacokinetics of Three SC Olanzapine Extended-release Formulations With Different Release Rates Following Single Administration in Participants With Schizophrenia or Schizoaffective Disorder
Brief Title: Open-label Trial Characterizing the PK of 3 SC Olanzapine Extended-release Formulations in Participants With Schizophrenia/Schizoaffective Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D LLC (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TV44749-NPC-10205
Record Dates: First submitted 2024-03-13; First posted 2024-03-19 (Actual); Results first posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia, Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Olanzapine (Fast-D) 425mg (Experimental): Single-dose injection
  Interventions: Drug: Olanzapine Extended Release
- Olanzapine (To-be-marketed) 425mg (Experimental): Single-dose injection
  Interventions: Drug: Olanzapine Extended Release
- Olanzapine (Slow-C) 425mg (Experimental): Single-dose injection
  Interventions: Drug: Olanzapine Extended Release
- ZYPREXA 5mg (Experimental): Single-dose injection
  Interventions: Drug: Olanzapine Immediate Release

INTERVENTIONS:
Drug: Olanzapine Extended Release — Powder and vehicle for injectable suspension
  Arms: Olanzapine (Fast-D) 425mg; Olanzapine (Slow-C) 425mg; Olanzapine (To-be-marketed) 425mg
Drug: Olanzapine Immediate Release — IntraMuscular Injection
  Other Names: ZYPREXA
  Arms: ZYPREXA 5mg

SUMMARY:
The primary objective of the study is to characterize the pharmacokinetics of 3 formulations of olanzapine.

A secondary objective is to evaluate the safety and tolerability of 3 formulations of olanzapine.

Another secondary objective is to characterize the pharmacokinetics of ZYPREXA.

The planned duration of the study for each participant is 19 weeks.

DETAILED DESCRIPTION:
All participants received immediate-release ZYPREXA and then were randomized into 1 of 3 extended-release olanzapine formulations.

ELIGIBILITY:
Inclusion Criteria:

* Body weight >50 kg and body mass index (BMI) within the range 18.5 to 38.0 kg/m2, inclusive, at the time of screening
* Agree to maintain current smoking or nonsmoking status at the time informed consent is obtained and throughout the trial until completion of the end of treatment or early termination (ET) visit (ie, nonsmoking participants must agree not to start smoking and participants who smoke will be excluded if they plan to discontinue smoking during the trial
* Agree to the inpatient periods required during the trial period
* Have a current confirmed diagnosis of schizophrenia or schizoaffective disorder according to an evaluation by the Investigator, using the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) (American Psychiatric Association 2013a)
* Have no ongoing or expected significant life events (eg, pending loss of housing, marital status change, long travel abroad, surgery) that could affect trial outcomes throughout the period of trial participation
* Women may be included only if they have a negative serum beta human chorionic gonadotropin (HCG) test result at screening; they are surgically sterile (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or postmenopausal
* Men must be sterile; or if they are potentially of reproductive competence and have sexual relationship with female partners of childbearing potential, they must use, together with their female partners, highly effective birth control methods for the duration of the trial and for 70 days after the last dose administration

NOTE- Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* Presence or have a history of clinically significant diseases of the renal, hepatic, gastrointestinal, cardiovascular, or musculoskeletal system, or presence or history of clinically significant immunological, endocrine, or metabolic diseases, neurological or psychiatric disorder(s) (other than schizophrenia)
* History or known risk of narrow-angle glaucoma
* Uncontrolled diabetes
* Major trauma or surgery in the 2 months before screening
* History of malignancy or treatment of malignancy in the last 5 years, excluding resected basal cell or squamous cell carcinoma of the skin
* The participant is a pregnant or lactating woman or plans to become pregnant during the trial or within 70 days after the last dose administration
* Personal or family history of arrhythmia, sudden unexplained death at a young age (before 40 years) in a first-degree relative, long QT syndrome, personal history of syncope, or history of uncontrolled high blood pressure

NOTE- Additional criteria apply, please contact the investigator for more information

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (5):
- United States (5):
  - Teva Investigational Site 15730, Los Alamitos, California
  - Teva Investigational Site 15727, Hollywood, Florida
  - Teva Investigational Site 15729, Atlanta, Georgia
  - Teva Investigational Site 15728, Decatur, Georgia
  - Teva Investigational Site 15726, Marlton, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be assessed for scientific merit, product approval status, and conflicts of interest. If the request is approved, patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please visit USMedInfo@tevapharm.com to make your request.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 183 participants signed the informed consent form for screening. Of these, 106 participants met eligibility criteria and were enrolled in the study. 91 participants were randomized to treatment arms.
Groups:
- ZYPREXA: Participants received a single injection of 5 milligrams (mg) of ZYPREXA, immediate-release solution, administered intramuscularly (IM) to the gluteal muscle.
- Cohort 1: Olanzapine (Fast-D): Participants received a single injection of 425 mg of olanzapine (Fast-D), extended-release formulation, administered subcutaneously (SC) to the abdomen.
- Cohort 2: Olanzapine (To-be-marketed): Participants received a single injection of 425 mg of olanzapine (To-be-marketed), extended-release formulation, administered SC to the abdomen.
- Cohort 3: Olanzapine (Slow-C): Participants received a single injection of 425 mg of olanzapine (Slow-C), extended-release formulation, administered SC to the abdomen.
Period: 1-Day Treatment Period
Arm/Group | ZYPREXA | Cohort 1: Olanzapine (Fast-D) | Cohort 2: Olanzapine (To-be-marketed) | Cohort 3: Olanzapine (Slow-C)
Started | 106 | 0 | 0 | 0
Received at Least 1 Dose of Study Drug | 98 | 0 | 0 | 0
Completed | 91 | 0 | 0 | 0
Not Completed | 15 | 0 | 0 | 0
Not completed — Enrolled But Not Treated | 8 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0
Not completed — Other Than Specified | 2 | 0 | 0 | 0
Period: 28-Day Treatment Period
Arm/Group | ZYPREXA | Cohort 1: Olanzapine (Fast-D) | Cohort 2: Olanzapine (To-be-marketed) | Cohort 3: Olanzapine (Slow-C)
Started | 0 | 29 | 31 | 31
Received at Least 1 Dose of Study Drug | 0 | 29 | 31 | 31
Completed | 0 | 28 | 29 | 31
Not Completed | 0 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0
Not completed — Other Than Specified | 0 | 1 | 0 | 0
Period: 8-Week Follow-up Period
Arm/Group | ZYPREXA | Cohort 1: Olanzapine (Fast-D) | Cohort 2: Olanzapine (To-be-marketed) | Cohort 3: Olanzapine (Slow-C)
Started | 0 | 28 | 29 | 31
Completed | 0 | 27 | 27 | 30
Not Completed | 0 | 1 | 2 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Other Than Specified | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Enrolled Analysis Set included all participants who signed an informed consent form (ICF) and were enrolled in the trial.
Groups:
- ZYPREXA Only (Not Randomized): Participants received a single injection of 5 mg of ZYPREXA, immediate-release solution, administered IM to the gluteal muscle.
- Cohort 1: Olanzapine (Fast-D): Participants received a single injection of 425 mg of olanzapine (Fast-D), extended-release formulation, administered SC to the abdomen.
- Total: Total of all reporting groups
Arm/Group | ZYPREXA Only (Not Randomized) | Cohort 1: Olanzapine (Fast-D) | Cohort 2: Olanzapine (To-be-marketed) | Cohort 3: Olanzapine (Slow-C) | Total
Number analyzed (Participants) | 15 | 29 | 31 | 31 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (11.95) | 45.7 (11.88) | 43.3 (11.39) | 42.1 (11.48) | 42.8 (11.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 11 | 6 | 10 | 29
  Male | 13 | 18 | 25 | 21 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 11 | 8 | 29
  Not Hispanic or Latino | 12 | 22 | 20 | 23 | 77
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 6 | 7 | 14 | 10 | 37
  Race: Black or African American | 9 | 22 | 14 | 19 | 64
  Race: Asian | 0 | 0 | 0 | 2 | 2
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Race: Other | 0 | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Olanzapine (Extended-release Formulation)
Time Frame: Randomization Day 1 to 84 days after randomization
Population: The Pharmacokinetic (PK) Analysis Set included all participants who had sufficient data to calculate at least 1 PK parameter for any of the olanzapine formulations (IM immediate release or SC extended release) and had no intercurrent events or deviations that affected the calculation of PK parameters. 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms (ng)/milliliter (mL)
Arm/Group | Cohort 1: Olanzapine (Fast-D) | Cohort 2: Olanzapine (To-be-marketed) | Cohort 3: Olanzapine (Slow-C)
Number analyzed (Participants) | 29 | 28 | 31
nanograms (ng)/milliliter (mL) | 39.26 (45.10) | 35.62 (67.55) | 29.68 (50.13)

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Study Drug Administration to the Last Measurable Concentration (AUC0-t) of Olanzapine (Extended-release Formulation)
Time Frame: Randomization Day 1 to 84 days after randomization
Population: The PK Analysis Set included all participants who had sufficient data to calculate at least 1 PK parameter for any of the olanzapine formulations (IM immediate release or SC extended release) and had no intercurrent events or deviations that affected the calculation of PK parameters. 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | Cohort 1: Olanzapine (Fast-D) | Cohort 2: Olanzapine (To-be-marketed) | Cohort 3: Olanzapine (Slow-C)
Number analyzed (Participants) | 27 | 26 | 30
hours*ng/mL | 20994.08 (33.77) | 20185.90 (47.35) | 18461.94 (35.44)

3. Primary Outcome: Area Under the Plasma Concentration-time Curve Extrapolated to Infinity (AUC0-inf) of Olanzapine (Extended-release Formulation)
Time Frame: Randomization Day 1 to 84 days after randomization
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | Cohort 1: Olanzapine (Fast-D) | Cohort 2: Olanzapine (To-be-marketed) | Cohort 3: Olanzapine (Slow-C)
Number analyzed (Participants) | 24 | 23 | 27
hours*ng/mL | 21703.07 (35.06) | 22146.09 (42.77) | 19011.66 (37.21)

4. Secondary Outcome: Number of Participants With at Least 1 Treatment-emergent Adverse Event (TEAE) Over the 28-day Period Following Administration of 1 of the SC Olanzapine Formulations
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who received the study drug without regard to possibility of causal relationship. A TEAE was defined as an AE that occurred after the first dose of study drug administration through the end of trial. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in the Reported AE section.
Time Frame: Randomization Day 1 through Randomization Day 29
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug (ZYPREXA IM or one of the Olanzapine SC extended-release formulations). This outcome measure reports data for the participants who received one of the Olanzapine SC extended-release formulations only.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Olanzapine (Fast-D) | Cohort 2: Olanzapine (To-be-marketed) | Cohort 3: Olanzapine (Slow-C)
Number analyzed (Participants) | 29 | 31 | 31
Participants | 9 | 12 | 9

5. Secondary Outcome: Number of Participants With at Least 1 Serious Adverse Event (SAE) Over the 28-day Period Following Administration of 1 of the SC Olanzapine Formulations
Description: The SAEs were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in the Reported AE section.
Time Frame: Randomization Day 1 through Randomization Day 29
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Olanzapine (Fast-D) | Cohort 2: Olanzapine (To-be-marketed) | Cohort 3: Olanzapine (Slow-C)
Number analyzed (Participants) | 29 | 31 | 31
Participants | 0 | 1 | 0

6. Secondary Outcome: Cmax of ZYPREXA (Immediate-release Formulation)
Time Frame: Up to 24 hours after administration of ZYPREXA (Day 4)
Population: The PK Analysis Set included all participants who had sufficient data to calculate at least 1 PK parameter for any of the olanzapine formulations (IM immediate release or SC extended release) and had no intercurrent events or deviations that affected the calculation of PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- ZYPREXA: Participants received a single injection of 5 mg of ZYPREXA, immediate-release solution, administered IM to the gluteal muscle.
Arm/Group | ZYPREXA
Number analyzed (Participants) | 97
ng/mL | 11.09 (82.89)

7. Secondary Outcome: AUC0-t of ZYPREXA (Immediate-release Formulation)
Time Frame: Predose (Day 4) up to 216 hours after administration of ZYPREXA (Day 13)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | ZYPREXA
Number analyzed (Participants) | 91
hours*ng/mL | 264.22 (48.14)

8. Secondary Outcome: Apparent Plasma Terminal Elimination Rate Constant (λz) of ZYPREXA (Immediate-release Formulation)
Time Frame: Predose (Day 4) up to 216 hours after administration of ZYPREXA (Day 13)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | ZYPREXA
Number analyzed (Participants) | 93
1/hour | 0.0159 (0.00381)

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 84
Description: All-cause mortality data were collected and reported for all enrolled participants; and Serious and Non-serious adverse events data were collected and reported for all participants who received at least 1 dose of study drug (ZYPREXA IM or one of the Olanzapine SC extended-release formulations).
Arm/Group | ZYPREXA | Cohort 1: Olanzapine (Fast-D) | Cohort 2: Olanzapine (To-be-marketed) | Cohort 3: Olanzapine (Slow-C)
All-Cause Mortality (participants affected / at risk) | 0/106 | 0/29 | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/29 | 1/31 | 0/31
Other Adverse Events (participants affected / at risk) | 18/98 | 8/29 | 11/31 | 6/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZYPREXA (N=98) | Cohort 1: Olanzapine (Fast-D) (N=29) | Cohort 2: Olanzapine (To-be-marketed) (N=31) | Cohort 3: Olanzapine (Slow-C) (N=31)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZYPREXA (N=98) | Cohort 1: Olanzapine (Fast-D) (N=29) | Cohort 2: Olanzapine (To-be-marketed) (N=31) | Cohort 3: Olanzapine (Slow-C) (N=31)
Injection site irritation (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (5) | 0 (0) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 6 (8) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 5 (5) | 1 (1) | 3 (3) | 2 (2)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2024-05-11): https://cdn.clinicaltrials.gov/large-docs/70/NCT06319170/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-11): https://cdn.clinicaltrials.gov/large-docs/70/NCT06319170/SAP_001.pdf